CLINICAL TRIAL: NCT01306344
Title: Qualitative Descriptive Study of the Meaning of the Ward Round
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo University College (Other)
Responsible Party: Stab forskning, innovasjon og utdanning, Oslo University Hospital
Other Study IDs: 2010/2607(REK)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Teaching Rounds
Keywords: Qualitative Research; Interview, Psychological; Patients; Nurses; Physicians

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients: Heterogeneous groups of patients (age, gender)
- Nurses: Heterogeneous groups of nurses (age, gender, working experience)
- Physicians: Heterogeneous groups of physicians (age, gender, working experience)

SUMMARY:
1. A qualitative descriptive design.
2. A phenomenologic approach to investigate the meaning of the ward round.
3. Interviews of patients, nurses and physicians.
4. A Master thesis.

ELIGIBILITY:
Inclusion Criteria:

* Grown-ups, normal cognitive function, speaks norwegian.

Exclusion Criteria:

* Children, vulnerable patientgroups, students.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients at a hospital ward. Nurses and physicians working at the same hospital ward. Heterogeneous groups.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-03 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bjorg Christiansen, PhD, Study Director — Oslo University College
Locations (1):
- Oslo University Hospital, Oslo, Norway